CLINICAL TRIAL: NCT04841187
Title: French Registry of Patients Initiating Systemic Treatment for Cutaneous Psoriasis
Brief Title: Assessing the Long Term Effectiveness and Safety of Systemic Treatments in Cutaneous Psoriasis
Acronym: PSOBIOTEQ
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201153; 2020-A03437-32 (Registry Identifier: Number ID-RCB)
Record Dates: First submitted 2021-03-08; First posted 2021-04-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; Adult; Systemic treatment; Biological therapy; Biosimilar therapy; small-molecule inhibitor of phosphodiesterase 4 (PDE4); Methotrexate; Ciclosporin
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PSOBIOTEQ is a national multicentric prospective non interventional study which aims to constitute a French registry of cutaneous psoriasis patients initiating systemic treatment (excluding acitretin and phototherapy) for moderate to severe cutaneous psoriasis. The general objective of PSOBIOTEQ registry is to describe the use, benefits and risks of conventional, biological, biosimilar and small-molecule inhibitor of phosphodiesterase 4 (PDE4) systemic treatments in a real-life setting.

The registry aims to meet many specific objectives and to fulfill ancillary studies. The PSOBIOTEQ registry concerns a largely similar population and has same objectives than the PSOBIOTEQ Cohort (NCT01617018). Indeed, data from the PSOBIOTEQ cohort will constitute the historical part of the registry and the cohort patients will pursue their follow-up in the registry framework, in order to enrich their follow up with new collected data.

DETAILED DESCRIPTION:
PSOBIOTEQ is a national multicentric prospective non interventional study which aims to constitute a French registry of cutaneous psoriasis patients initiating systemic treatment (excluding acitretin and phototherapy) for moderate to severe cutaneous psoriasis.

The exposure of interest is the exposure to any major systemic treatment (excluding acitretin and phototherapy) for moderate to severe cutaneous psoriasis and marketed in France at the time of inclusion of the patient in the registry.

The nature of the systemic treatment as well as its administration modalities are defined by the investigator according to usual practice.

The dermatology departments participating to the PSOBIOTEQ cohort were solicited for participation to the PSOBIOTEQ registry.

The PSOBIOTEQ registry will start in 2020 with 28 dermatology departments. The PSOBIOTEQ cohort started in 2012 and was finalized in 2020. The PSOBIOTEQ registry continues from 2020 till 2025.

The inclusion will last 4 years with a follow-up of at least 1 year of the latest patient and until the end of the research for the other patients with a 6 month periodicity and at least one visit per year, for the data collection (complying with good clinical practice for these patients). Each included patient remains followed-up as long as he doesn't object.

All data required will be collected and registered in a single database (eCRF). The statistical analyses planned in the research protocol and those responding to requests for additional data from the Transparency Committee in the context of the provision of biomedicines, their biosimilars or other major systemic treatments obtaining Marketing Authorization in the treatment of cutaneous psoriasis, will be performed by the pharmaco-epidemiology center (CEPHEPI) under the responsibility of Pr Florence TUBACH of La Pitié Salpêtrière hospital.

The ancillary studies analyses responding to general objectives of the registry dealing with psoriasis and its course, the terms of use or the benefits and risks of its treatments (for example in case of identification of safety signals) or new research questions emerging during the conduct of the study (or after the study), whose realization is validated by the scientific committee of the registry may be carried out by CEPHEPI or the academic teams participating in the PSOBIOTEQ registry.

A calculation of the sample size is not justified for this study as it aims to describe all the patients initiating systemic treatment for cutaneous psoriasis in the participating centers. However, based on the rate of inclusion in the PSOBIOTEQ cohort, an inclusion rate of 500 patients per year can be estimated (therefore 2000 patients to be included in 4 years).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Had been informed about the objectives and progress of the research, and not opposed to the collection of his data
* Consulting or hospitalized in one of the departments participating in the study :
* For a cutaneous psoriasis (clinical diagnosis)
* And at least one of the two criteria below must be met :

  * In whom a systemic treatment is initiated (excluding phototherapy or acitretin) that he has never received in the past * (a patient who has already received a biomedicine (princeps and / or biosimilar (s)) in the past cannot be included under the same biomedicine (princeps and / or biosimilar (s)). Patients initiating treatment with methotrexate or ciclosporin must be naïve of any biomedicine.
  * Patients included in the PSOBIOTEQ 1 cohort

Exclusion Criteria:

* Patient for whom cutaneous psoriasis is not the main reason for systemic treatment (psoriatic arthritis, or concomitant Crohn's disease, etc.);
* Patient unable to comply with the registry's follow-up procedures (not reachable by phone, unable to complete the self-questionnaire) or whose monitoring is deemed difficult;
* Patient for whom the treatment administered at inclusion cannot be identified (patient included in a randomized double-blind biomedicine research protocol, for example).
* Patient under guardianship or curatorship

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied population corresponds to adult patients initiating systemic treatment (excluding acitretin and phototherapy) for moderate to severe cutaneous psoriasis in the centers participating to the PSOBIOTEQ Registry.
  The PSOBIOTEQ registry concerns a largely similar population and has same objectives than the PSOBIOTEQ Cohort (NCT01617018). Indeed, data from the PSOBIOTEQ cohort will constitute the historical part of the registry and the cohort patients will pursue their follow-up in the registry framework, in order to enrich their follow up with new collected data.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of skin cancer | Up to 5 years of follow up for each patient
  Occurrence of skin cancer (spinocellular carcinomas [including carcinoma in situ (Bowen) and keratoacanthomas], basocellular carcinomas and melanomas).

SECONDARY OUTCOMES:
Physicians global assessment of disease (PGA) score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Psoriasis Area and Severity Index (PASI) Score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Body surface area | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Dermatology Life Quality Index (DLQI) Score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Global Self Assessed (GSA) Score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
EuroQol 5-Dimension Health Status Questionnaire (EQ-5D) index score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Patient Report of Extent of Psoriasis Involvement (PREPI) score | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients reporting acceptable symptom state : acceptance to remain for the rest of their lives with the level of disease activity they had during the last 48 hours | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients reporting clinically important improvement in psoriasis activity during the last 48 hours compared to baseline | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Occurrence of Adverse Events and Serious Adverse Events | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Occurrence of Events of special interest such as infectious diseases, autoimmune diseases, lymphoma and blood disorders, multiple solid tumors, cardiovascular diseases, etc. | [Time Frame: Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Drug survival rate (proportion of patients still exposed to treatment | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Socio-demographic and clinical data: age, sex, socio-professional category, body mass index (BMI) and phototype (Fitzpatrick) | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Lifestyle data: family life, tobacco consumption, alcohol consumption and history of natural and artificial UV exposure | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients with history and comorbidities | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients with previous systemic treatments including phototherapy and acitretin | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients with systemic treatments | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Number of patients with concomitant treatments | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Daily dose of systemic treatments | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.
Therapeutic strategy: duration of systemic treatments, dosages, change in systemic treatments, reasons for modifications of systemic treatments | Each patient will be followed for at least 1 year (The duration of follow-up is 5 years), data being collected at each visit (approximately every 6 month) with a minimum of one medical visit per year.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSIDOW, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: Yes
Undecided